CLINICAL TRIAL: NCT06104709
Title: Local and Peripheral Immune Responsive Landscape Induced by Local Cryoablation in Patients With Lung Adenocarcinoma
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: China-Japan Friendship Hospital (Other)
Responsible Party: Principal Investigator, Gang Hou, Principle Investigator, China-Japan Friendship Hospital
Other Study IDs: ZRJY2021-BJ08-02-06
Record Dates: First submitted 2023-10-24; First posted 2023-10-27 (Actual); Last update posted 2023-10-27 (Actual); Status verified 2023-10

CONDITIONS: Lung Adenocarcinoma; Local Cryoablation
Keywords: Lung Adenocarcinoma; local cryoablation; immune landscape; metabolic changes
MeSH Terms: conditions — Adenocarcinoma of Lung

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- LUAD patients undergoing cryoablation: No interventions.

SUMMARY:
The goal of this observational study is to learn about local and peripheral immune and metabolic changes in patients with lung adenocarcinoma undergoing cryoablation. The main question it aims to answer are:

* local and peripheral immune changes in patients with lung adenocarcinoma undergoing cryoablation.
* local and peripheral metabolic changes in patients with lung adenocarcinoma undergoing cryoablation.

Peripheral blood, biopsy tissues of patients will be collected at the baseline and after cryoablation. Single-cell sequencing, single-cell immune bank, metabolomics and spatial metabolomics will be used to explore the local and peripheral immune changes and metabolites changes in patients with lung adenocarcinoma before and after cryoablation.

ELIGIBILITY:
Inclusion Criteria:

1. Primary or metastatic lung cancer with definite pathological diagnosis.
2. Patients are not suitable for thoracotomy due to serious lung or systemic disease.
3. Peripheral lung cancer involves pleura and chest wall, which cannot be completely removed by surgical resection.
4. There are indications for surgical resection, but the patient refuses surgery.
5. Single tumor, maximum diameter ≤5cm; Or the number of tumors ≤3, the maximum diameter ≤3cm.
6. ECOG-PS score≤2.
7. Patients with an expected survival of more than three months.
8. Patients have not participated in other clinical validation within 3 months.
9. Subjects voluntarily sign informed consent.

Exclusion Criteria:

1. Serious heart and brain disease or other mental illness.
2. Severe pulmonary fibrosis, especially drug-induced pulmonary fibrosis.
3. Patients with previous severe pulmonary dysfunction, pulmonary ventilation disorder, and multiple pulmonary bulla.
4. A history of immunodeficiency, including a positive HIV test (enzyme-linked immunoassay and Western spot assay).
5. Patients treated with chemotherapy, radiotherapy, interventional therapy, ablative therapy or surgery within 30 days before surgical treatment.
6. There is a serious bleeding tendency, platelets less than 50×109 /L and coagulation function is seriously disturbed.
7. Coagulation index (PT, TT, APTT) > 2.5 times the upper limit of normal.
8. Ablation of ipsilateral malignant pleural effusion is not well controlled.
9. Poor general condition, multiple organ failure, cachexia, severe anemia and nutritional metabolism disorders.
10. Patients with extensive extrapulmonary metastasis are not suitable for ablative therapy.
11. People who regularly use sedatives, sleeping pills, tranquilizers or other addictive drugs.
12. Pregnant or breastfeeding women.
13. Patients who cannot evaluate the efficacy.
14. Other conditions determined by the investigators to be unsuitable for inclusion, such as inability to tolerate cryoablation surgery, difficulty in follow-up, and other serious diseases.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with lung adenocarcinoma who have indictions of local cryoablation without any other contraindications.
Sampling Method: Non-Probability Sample
Enrollment: 10 (Estimated)
Dates: Start 2023-12-01 (Estimated); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
cryoablation completion | 1 month
  patients complete local cryoablation